CLINICAL TRIAL: NCT05372900
Title: Nutritional Intervention to Improve Sleep Quality and Improve Next-day Mood and Cognitive Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 21.03.DAI
Record Dates: First submitted 2021-12-02; First posted 2022-05-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Sleep
Keywords: Subjective sleep complaints
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a double-blind, controlled, randomized, 2-arm, cross-over, group sequential design clinical trial. Subjects will receive the two different interventions in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - Control product (Experimental): Subject will start with consuming the test product daily for total 14 days (during intervention 1 period). After the 4 - 6 weeks wash out, subject will then consume the control product daily for total 14 days (during intervention period 2).
  Interventions: Other: Test Product; Other: Control Product
- Control - Test product (Experimental): Subject will start with consuming the control product daily for total 14 days (during intervention 1 period). After the 4 - 6 weeks wash out, subject will then consume the test product daily for total 14 days (during intervention period 2).
  Interventions: Other: Test Product; Other: Control Product

INTERVENTIONS:
Other: Test Product — Whey Protein Isolate with Mulberry leaf extract
Other: Control Product — Wheat Protein Hydrolysate

SUMMARY:
The study aim to test the effect of a meal complement to be taken in combination with an evening meal with a glycemic load of 55, to improve sleep quality.

DETAILED DESCRIPTION:
Considering emerging evidence on the role of the macro and micro-nutrient composition of evening meals, the intervention used in this study will be designed to provide the necessary nutrients to promote sleep quality. The IP will be a low caloric nutritional solution, combining:

* Ingredients lowering glycemic response to evening meals to promote sleep quality
* a protein source rich in bioavailable tryptophan to promote sleep quality
* supporting ingredients contributing to sleep initiation

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able provide written informed consent (in English)
2. Aged 25-50
3. BMI range from 18.5 to 24.9 kg/m2
4. Subjective sleep complaints (PSQI > 5)

Exclusion Criteria:

1. Diagnosed food allergy or other intolerance to the investigational products, control products and standardized meals
2. Significant past medical and psychiatric history and ongoing chronic conditions for example cardiovascular disease, respiratory disease, metabolic disorder, endocrine disorder (e.g. diabetes mellitus, history of hypoglycemia), and neurological and psychiatric conditions, and conditions that the investigator deem inappropriate to enter the clinical trials
3. Significant medication history including use of corticosteroid in oral or systemic format and antidepressants (e.g. Selective Serotonin Reuptake Inhibitors, Monoamine Oxidase Inhibitors)
4. Pregnant or intending to conceive during the course of clinical trial and up to one month after trial conclusion, or not able to comply with a highly effective form of birth control or lactating during the clinical trial. Highly effective contraception includes hormonal methods, such as the contraceptive pill or implant, or an intrauterine device (IUD), or barrier methods such as diaphragm plus spermicide or condom plus spermicide. Pregnancy status will be assessed using urinary dipsticks at the beginning and end of the study period (V0 and V9).
5. Parents of children less than 12 months of age, which is a known factor of sleep disturbances.
6. Peri- and post-menopausal women
7. Known or diagnosed sleep disorders
8. Special diets, including for instance halal food preference, vegetarian, high protein or weight loss program, and diets with either too low (< 35% daily energy from CHO; e.g., ketogenic diet, Atkins diet, zero-carb diet, low-carb paleo/Mediterranean diet, carb cycling diet) or too high carbohydrate (>70% daily energy from CHO) content .
9. Chronic exercisers, defined as subjects exercising > 1 h/day for at least 5 days/week
10. Caffeine consumption over the recommended daily limit (above 400 mg; equivalent to approximately 4-5 cups of coffee)
11. Substance abuse including over the limit alcohol consumption (2 standard drinks/day for males, 1 standard drink/day for female)
12. Cigarette and Tobacco Smokers
13. Intake of dietary supplements that may affect sleep conditions (e.g. melatonin, theanine, tryptophan, GABA, magnesium, zinc)
14. Subjects not willing and/or not able to comply with scheduled visits and the requirements of the study protocol.
15. Participating in other clinical trials or had been participating in other clinical trial in the preceding 1 month.
16. Subjects belonging to a household where at least one other person is taking part in the trial.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Changes in sleep efficiency (actigraphy) | Day 1 (V1) to Day 15 (V2), Day 22 (V3) to Day 37, Day 38 (V5) to Day 45, Day 59 (V6) to Day 65, Day 66 (V7) to Day 79, Day 80 (V8) to Day 87 (V9)
  Calculated as '(total time asleep / time in bed) X 100; sleep efficiency above 85% is considered good.
Change in sleep latency (actigraphy) | Day 1 (V1) to Day 15 (V2), Day 22 (V3) to Day 37, Day 38 (V5) to Day 45, Day 59 (V6) to Day 65, Day 66 (V7) to Day 79, Day 80 (V8) to Day 87 (V9)
  Measured as the amount of time it takes subjects to fall asleep after going to bed (in minutes)

SECONDARY OUTCOMES:
Changes in self-reported sleep quality via Actigraphy | Day 1 (V1) to Day 15 (V2) , Day 22 (V3) to Day 37, Day 38 (V5) to Day 45, Day 59 (V6) to Day 65, Day 66 (V7) to Day 79, Day 80 (V8) to Day 87 (V9)
  Changes in WASO & total sleep duration
Changes in self-reported sleep quality via KSD | Day 1 (V1), Day 15 (V2), Day 22 (V3), Day 23, Day 24 (V4) to Day 37, Day 45 and 65, Day 66 (V7) to Day 79, Day 87 (V9)
  Changes in self-reported sleep quality measured through questionnaire Karolinska Sleep Diary (KSD)
Changes in self-reported sleep quality via ESS | Day 1 (V1) & Day 15 (V2), Day 23, 31, 37, 45, 65, 73, 79, 87)
  Changes in self-reported sleep quality measured through questionnaire Epworth Sleepiness Scale (ESS)
Glycemia | Day 1 (V1) to Day 14, Day 24 (V4) to Day 37, Day 66 (V7) 7 to Day 79
  Glycemia measured by continuous glucose monitoring:
  * Glucose response of the evening standard meal with the test product or the control product
  * Glucose excursion during the night (from time to bed to wakening)
  * Subsequent breakfast
Mood states, alertness, and sleepiness via BMIS | Day 22 (V3), Day 23 to Day 37, Day 65, Day 66 (V7) to Day 79
  Questionnaire Brief Mood Introspection Scale (BMIS)
Mood states, alertness, and sleepiness via KSS | Day 22 (V3), Day 23 to Day 37, Day 65, Day 66 (V7) to Day 79
  Questionnaire Karolinska Sleepiness Scale (KSS)
Mood states, alertness, and sleepiness via POMS-SF 2 | Day 22 (V3), Day 23, 31, 37, 65, 73, 79
  Questionnaire Profile of Mood States - Short Form 2 (POMS-SF 2)
Cognition tasks via Immediate & delayed free recall | Day 22 (V3), Day 23, 37, 65, 79
  Immediate & delayed free recall
Cognition task PVT | Day 22 (V3), Day 23, 31, 37, 65, 73, 79
  Psychomotor Vigilance Task (PVT)
Cognition test N-back task | Day 22 (V3), Day 23, 31, 37, 65, 73, 79
  N-back task
Cognition test Go/No-Go task | Day 22 (V3), Day 23, 31, 37, 65, 73, 79
  Go/No-Go task
Cognition task NASA-TLX | Day 22 (V3), Day 23, 31, 37, 65, 73, 79
  NASA task load index (NASA-TLX)

OTHER OUTCOMES:
Cortisol levels in the morning | Day 24 (V4), Day 28 (V5), Day 66 (V7), Day 80 (V8)
  Cortisol levels in saliva as an objective index of stress
Melatonin synthesis marker (6-sulfatoxymelatonin) | Day 24 (V4), Day 28 (V5), Day 66 (V7), Day 80 (V8)
  6-sulfatoxymelatonin levels in urine as an index of melatonin synthesis, which will be reported as a ratio of urinary 6-sulfatoxymelatonin to urinary creatinine.
Assess effect of sleep hygiene behaviors and life events on sleep patterns | Visit 0 (pre Day1), Day 23, Day 65
  Sleep hygiene questionnaire
Change in sleep efficiency, calculated as '(total time asleep / time in bed) X 100; sleep efficiency above 85% is considered good | Day 1 (V1) to Day 15 (V2), Day 22 (V3) to Day 37, Day 38 (V5) to Day 45, Day 59 (V6) to Day 65, Day 66 (V7) to Day 79, Day 80 (V8) to Day 87 (V9)
  Measure of sleep parameter using the commercial sensor Oura ring
Change in sleep latency (mins), measured in time needed to fall asleep after going to bed. | Day 1 (V1) to Day 15 (V2), Day 22 (V3) to Day 37, Day 38 (V5) to Day 45, Day 59 (V6) to Day 65, Day 66 (V7) to Day 79, Day 80 (V8) to Day 87 (V9)
  Measure of sleep parameter using the commercial sensor Oura ring
Change in WASO (actigraphy) - proportion of people reaching < 30 mins | Day 1 (V1) to Day 15 (V2), Day 22 (V3) to Day 37, Day 38 (V5) to Day 45, Day 59 (V6) to Day 65, Day 66 (V7) to Day 79, Day 80 (V8) to Day 87 (V9)
  Measure of sleep parameter using the commercial sensor Oura ring
Change in total sleep duration (mins; actigraphy) | Day 1 (V1) to Day 15 (V2), Day 22 (V3) to Day 37, Day 38 (V5) to Day 45, Day 59 (V6) to Day 65, Day 66 (V7) to Day 79, Day 80 (V8) to Day 87 (V9)
  Measure of sleep parameter using the commercial sensor Oura ring.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chee, Principal Investigator — National University of Singapore
Locations (1):
- Centre for Sleep and Cognition, NUS Yong Loo Lin School of Medicine, Singapore, Singapore

REFERENCES:
- [Derived] Soon CS, Thota R, Owen L, Tian L, Martin FP, Mantantzis K, Cherta-Murillo A, Campos VC, Chkroun C, Lavalle L, Hartweg M, St-Onge MP, Chee MWL, Darimont C. Mulberry leaf extract combined with tryptophan improves sleep and post wake mood in adults with sleep complaints - A randomized cross-over study. Eur J Nutr. 2025 Mar 12;64(3):124. doi: 10.1007/s00394-025-03643-8. PMID 40072601